CLINICAL TRIAL: NCT01912547
Title: Thromboelastography During Surgery for Malignant Pleural Mesothelioma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ju-Mei Ng, Instructor of Anaesthesia, Brigham and Women's Hospital
Other Study IDs: 2013P000653
Record Dates: First submitted 2013-07-27; First posted 2013-07-31 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Coagulopathy; Mesothelioma
MeSH Terms: conditions — Hemostatic Disorders; Mesothelioma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Blood draw for TEG analysis: TEG analysis of blood from patients at different points in time
  Interventions: Procedure: Blood draw for TEG analysis

INTERVENTIONS:
Procedure: Blood draw for TEG analysis — Blood drawn for TEG analysis

SUMMARY:
Surgery for malignant pleural mesothelioma is complex and prolonged, and may involve significant blood loss with considerable blood and product transfusion. Thromboelastography (TEG) is a global assay of coagulation that uses whole blood to produce a tracing that records kinetic changes in clot formation. This study aims provide a better understanding of the coagulation profile of these patients, and will form the basis of a TEG-based transfusion algorithm for future surgeries for mesothelioma.

DETAILED DESCRIPTION:
Thromboelastography can provide more in-depth and quicker analysis of the complex coagulation processes during surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients undergoing elective surgery for malignant pleural mesothelioma

Exclusion Criteria:

* Unwilling or unable to provide consent
* History of bleeding disorder
* On medications that may affect hemostasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing surgery for malignant pleural mesothelioma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Coagulation profile during extrapleural pneumonectomy or pleurectomy | Surgical period (4-6 hours)
  Reaction time, alpha angle, maximum amplitude and clot lysis from thromboelastography give a better picture of coagulation at different phases of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Mei Ng, MD, Principal Investigator — BWH
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States